CLINICAL TRIAL: NCT06786741
Title: Culturally Responsive Intervention Incorporating AI to Promote Healthy Integration Among Afghan Evacuees in Illinois and Tennessee (Pilot Study)
Brief Title: Afghan Evacuee Resettlement for Stronger Communities (AER)
Acronym: AER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Project# 3964
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Stress Reduction; Healthy Relationships; Emotional Wellbeing
Keywords: evacuees; Afghan; stress; culturally responsive; integration
MeSH Terms: interventions — Aerosols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AER Intervention (Experimental): Intervention participants are provided with a 3 week rapid intervention.
  Interventions: Behavioral: AER for Stronger Communities
- Control (Placebo Comparator): Control participants are provided access to short videos across the same 3 week period.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Behavioral: AER for Stronger Communities — 3 week rapid intervention aimed at reducing stress.
  Arms: AER Intervention
Other: Placebo Comparator — 3 week short video program (control)
  Arms: Control

SUMMARY:
Background. Under Operation Allies Welcome, approximately 88,500 Afghan evacuees have resettled in the United States (US). Evacuees face unique integration, well-being, and mental health challenges. Settlement is nationwide, including key locations of Illinois (IL) and Tennessee (TN).

Study aims. In the proposed study, investigators will pilot test a 3-week culturally responsive and flexible, sprint (rapid) intervention, AER (Afghan Evacuee Resettlement) for Stronger Communities, with Afghan evacuees in IL and TN. A beta version of the first-ever AI platform, Dost, for Afghan evacuees will also be tested. Innovation. This is the first flexible and culturally responsive intervention and AI app created for Afghan evacuees to be delivered in English and Dari.

Up-to-date data from evacuees over the past year inform this intervention. Methods. To pilot test the intervention, a randomized control trial (RCT) with an optional waitlist will be conducted with approx. 50-60 evacuees across IL and TN. Community liaisons from partner agencies will also be recruited for intervention delivery. Participants in the intervention group will also be able to access the AI platform. Evacuees and liaisons will be invited to provide feedback on the intervention and evacuees will be invited to provide feedback on the platform. Expected results. Investigators expect to test the central hypothesis of the study, that individuals who receive the sprint intervention and access the AI platform will have reduced stress outcomes (integration, social relationships, and mental health) compared to those who do not. Impact. Findings will build new evidence for migrants in Chicago and nationally. This project will also further interdisciplinary collaboration across Loyola University Chicago and beyond.

DETAILED DESCRIPTION:
Background. Under Operation Allies Welcome, approximately 88,500 Afghan evacuees have resettled in the United States (US). Evacuees face unique integration, well-being, and mental health challenges. Settlement is nationwide, including key locations of Illinois (IL) and Tennessee (TN).

Study aims. In the proposed study, investigators will pilot test a 3-week culturally responsive and flexible, sprint (rapid) intervention, AER (Afghan Evacuee Resettlement) for Stronger Communities, with Afghan evacuees in IL and TN. A beta version of the first-ever AI platform, Dost, for Afghan evacuees will also be tested. Innovation. This is the first flexible and culturally responsive intervention and AI platform created for Afghan evacuees to be delivered in English and Dari.

Up-to-date data from evacuees over the past year inform this intervention. Methods. To pilot test the intervention, a randomized control trial (RCT) with an optional waitlist will be conducted with 50-60 evacuees across IL and TN. Community liaisons from partner agencies will also be recruited for intervention delivery. Participants in the intervention group will also be able to access the AI platform. Evacuees and liaisons will be invited to provide feedback on the intervention and evacuees will be invited to provide feedback on the platform. Expected results. Investigators expect to test the central hypothesis of the study, that individuals who receive the sprint intervention and access the AI platform will have reduced stress outcomes (integration, social relationships, and mental health) compared to those who do not. Impact. Findings will build new evidence for migrants in Chicago and nationally. This project will also further interdisciplinary collaboration across Loyola University Chicago and beyond.

The project is closely aligned with the priorities of the Schreiber Venture Fund that funded the pilot testing. Ultimately, findings will also lay the foundation for a future R01 NIH grant and have transdisciplinary implications.

ELIGIBILITY:
1. 18 years old or older, resettled to US post-2021 from Afghanistan
2. speaks English or Dari
3. has access to smart phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Stress reduction | Weeks 0, 1, 2,3, 4-week follow up
  Reduced stress as measured by PSS-4 instrument (0=never, 1=almost never, 2=sometimes, 3=fairly often, 4=very often
  *some scoring and questions were modified to make them culturally responsive.
Integration | Weeks 0, 1, 3, 4-week follow up
  IPL Integration Index (1 to 5, 1 low, and 5 is high); Economic self-efficacy (1=strongly disagree, 2=disagree, 3=neutral, 3=agree, 5=strongly agree)
  *some scoring and questions were modified to make them culturally responsive.
Healthy Relationships | Weeks 0, 2, 3, 4-week follow up
  Healthy relationships as measured by Relationship Assessment Scale (1=low, 2, 3, 4, 5=high); Brief Family Relationship Scale (1=strongly disagree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree); Gender role beliefs scale (1=strongly agree, 2=moderately agree, 3=slightly agree, 4=undecided, 5=slightly disagree, 6=moderately disagree, 7=strongly disagree.
  *some scoring and questions were modified to make them culturally responsive.
Emotional Wellbeing | Weeks 0, 3, 4-week follow up
  Emotional wellbeing as measured by Post-migration stress scale (1=never, 2=seldom, 3=sometimes, 4=often, 5=very often), brief Cope inventory (1=haven't been doing this at all, 2=been doing a little bit, 3=doing this a medium amount, 4=doing this a lot)
  *some scoring and questions were modified to make them culturally responsive.
Psychological distress | Weeks 0, 1, 2,3, 4-week follow up
  Kessler-6 to measure psychological distress (1=all of the time, 2=most of the time, 3=some of the time, 4=a little of the time, 5=none of the time)
  *some scoring and questions were modified to make them culturally responsive.

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided